CLINICAL TRIAL: NCT06348459
Title: Registry of Catheter Intervention in Pulmonary Embolism
Acronym: RiTEP
Status: Recruiting | Type: Observational
Sponsor: Hospital San Carlos, Madrid (Other)
Collaborators: Asociación de Cardiología Intervencionista de la Sociedad Española de Cardiología (Unknown)
Responsible Party: Principal Investigator, Pablo Salinas, MD, PhD, Hospital San Carlos, Madrid
Other Study IDs: 18/010-E
Record Dates: First submitted 2023-11-09; First posted 2024-04-04 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Pulmonary Embolism; Pulmonary Embolism Acute Massive; Pulmonary Embolism Acute; Pulmonary Embolism and Thrombosis; Pulmonary Thromboembolisms
Keywords: Aspiration Thrombectomy; Percutaneous Aspiration Thrombectomy; Local Thrombolysis
MeSH Terms: conditions — Pulmonary Embolism; Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Multicenter longitudinal observational ambispective (retrospective cases from 2014 and prospective from 2018 onwards) cohort study. The registry recruits a series of consecutive patients admitted for moderate-high risk or high-risk pulmonary embolism (according to 2019 European Society of Cardiology guidelines) treated invasively. This study aims to describe the acute management of the safety and effectiveness of different percutaneous interventions for acute pulmonary embolism.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (aged 18 years old or older)
* confirmed diagnosis of acute PE (on computed tomography or echocardiogram plus pulmonary angiography)
* high-risk PE or intermediate-high risk according to ESC risk stratification in the 2019 guidelines (briefly, elevated cardiac biomarkers [troponin or N-terminal pro-B-type natriuretic peptide], and right ventricle to left ventricle ratio > 0.9 [on computed tomography or echocardiogram], and PE severity index III to IV or simplified PE severity index=1
* eligibility for catheter-directed intervention

Exclusion Criteria:

* unconfirmed diagnosis of PE
* undefined risk stratification, and
* PE with uncertain chronology or beyond seven days of symptom initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients admitted for moderate-high risk or high-risk PE and treated invasively with any kind of catheter-directed intervention.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-18 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
All cause-death | during hospital admission (up to day 10)

SECONDARY OUTCOMES:
all cause-death | 48 hours
all cause-death | 30 days
all cause-death | 2 year
procedural success | 48 hours
  defined as technical procedure completed without procedural complications or 48-hour death
in-hospital complications | during hospital admission (up to day 10)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinico San Carlos, Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ramos-Lopez N, Ferrera C, Luque T, Enriquez-Vazquez D, Mahia-Casado P, Galvan-Herraez L, Pedrajas JM, Salinas P; working group. Impact of a pulmonary embolism response team initiative on hospital mortality of patients with bilateral pulmonary embolism. Med Clin (Barc). 2023 Jun 9;160(11):469-475. doi: 10.1016/j.medcli.2022.12.017. Epub 2023 Feb 16. English, Spanish. PMID 36801109
- [Background] Salinas P, Vazquez-Alvarez ME, Salvatella N, Ruiz Quevedo V, Velazquez Martin M, Valero E, Rumiz E, Jurado-Roman A, Lozano I, Gallardo F, Amat-Santos IJ, Lorenzo O, Portero Portaz JJ, Huanca M, Nombela-Franco L, Vaquerizo B, Ramallal Martinez R, Maneiro Melon NM, Sanchis J, Berenguer A, Gallardo-Lopez A, Gutierrez-Ibanes E, Mejia-Renteria H, Cordoba-Soriano JG, Jimenez-Mazuecos JM. Catheter-directed therapy for acute pulmonary embolism: results of a multicenter national registry. Rev Esp Cardiol (Engl Ed). 2024 Feb;77(2):138-147. doi: 10.1016/j.rec.2023.06.005. Epub 2023 Jun 22. English, Spanish. PMID 37354942